CLINICAL TRIAL: NCT05358067
Title: Predictability of the Clinical Global Impression Scale (CGI) in Post Immediate in Psychotraumatic Impact
Acronym: PRECLIP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Arras (Other)
Collaborators: F2RSM Psy (Hauts-de-France Regional Federation for Research in Psychiatry and Mental Health) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-02
Record Dates: First submitted 2022-04-11; First posted 2022-05-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate correlation between Clinical Global Impression Scale (CGI) score immediately in patients who have experienced psychotrauma and occurrence of posttraumatic stress disorder at distance from traumatic event. This could allow, in future, implementation of a systematic telephone reminder of psychotraumatized patients when they have a high score on the CGI scale, and thus detect onset of a stress disorder as early as possible, post-traumatic and orientation of these patients on specialized care.

DETAILED DESCRIPTION:
A functional unit of Urgent Medical Aid Service (SAMU), Medical-psychological emergency cell (CUMP) is an emergency medical device and provides immediate and post-immediate medico-psychological care for mentally injured people in psychotraumatic situations. CUMP also ensures immediate post follow-up of these patients, as well as departmental organization of psychotrauma consultation.

During the course of the treatment, victims are oriented, with a telephone callback which can be decided, allowing a remote reassessment of any psychotraumatic sequelae of the event. This phone reminder is part of routine practice following a CUMP intervention. The objective is then early detection of sequelae allowing rapid orientation on specific care pathways, in particular on the consultation of psychotrauma.

Post-traumatic stress disorder is a syndromic entity reactive to experience of a traumatogenic event (defined by the brutal, sudden and unexpected confrontation with death, or the loss of physical or psychological integrity), bringing together intrusive symptoms of reliving, behavioral avoidance of stimuli related to the traumatic event, persistent negative alterations in cognitions and mood, and neurovegetative hyperactivity, causing clinically significant distress and impaired the usual functioning of the subject.

Experiencing a psychotraumatic event in one's life is a frequent experience. Epidemiological data show a lifetime prevalence of around 30%. During and/or in the hours following a psychotraumatic event, people experience psychological, physiological and emotional upheavals called peritraumatic distress. Although most people recover on their own, a portion (8.3%) develop post-traumatic stress disorder.

However, one of the main characteristics of post-traumatic stress disorder is the presence of avoidance symptoms. Avoidance can take different forms such as non-confrontation with all the evocative clues of the traumatic event such as places, people and situations related to the traumatic event, but also the avoidance of thoughts, memories, conversations related to the traumatic event. This avoidance of thoughts and conversations can be a barrier to entry into trauma-focused psychotherapy. Indeed, talking about the traumatic event goes against this avoidance. A proactive approach at a distance from the event to re-evaluate the symptomatology of the people involved and thus propose an orientation towards specialized care in the field of psychotrauma in order to counter avoidance would seem entirely relevant.

Indeed, studies show the interest of a telephone follow-up by the Medical-Psychological Unit 15 days before an emergency repatriation of French people during the Lebanon war in 2016. On the one hand, remote telephone reminder of event is experienced positively by the people involved in the event and was able to highlight the presence of post-traumatic stress symptoms in 23% of cases. On the other hand, 56% of people were able to be referred to appropriate medio-psychological care following this telephone interview.

However, depending on the situation, all of the subjects involved in a psychotraumatic event cannot be reassessed, especially when event involves too many people. On the other hand, a significant proportion of subjects will not present psychotraumatic sequelae. Under these conditions, it seems appropriate to be able to define the proportion of psychotraumatized subjects most at risk of developing post-traumatic stress disorder (PTSD). Data from literature find that a high level of peritraumatic distress is largely associated with severity of post-traumatic stress symptoms .

Thus, peritraumatic distress reactions would be a good indicator of risk of developing a subsequent post-traumatic stress disorder. Several questionnaires exist to assess this peritraumatic distress. However, in a disaster situation and in view of the large number of victims potentially involved, it may be interesting to use a rapid and global assessment tool.

To do this, the severity item of the global clinical impression scale would respond to this clinical reality.

Research hypothesis

Hypothesis is that the severity item of the global clinical impression scale evaluated immediately after in a subject who has experienced a psychotraumatic event is a predictor of post-traumatic stress symptoms at 1 month and 6 months. Investigators expect a correlation between the scores of the PDI and the severity item of the global clinical impression while controlling the socio-demographic characteristics of the worker as well as his clinical experience. Patients included will have similar profiles and will be confronted with the same type of traumatic event.

Brief Protocol

* Inclusion visit : psychiatric assessment, socio-demographic data, questionnaire (CGI and Peritraumatic Distress Inventory scale(PDI))
* Follow-up visit: M1 and M6 : phone call (Post traumatic stress disorder Checklist Scale questionnaire (PCL 5), Mini International Neuropsychiatric Interview (MINI) : major depressive episod, alcohol consumption disorder, substance-related disorder (non-alcoholic).

Expected results

Investigators expect this work to confirm the prediction between the initial score on the CGI and the score at M1 and M6 on the PCL5. This result will make it possible to define an initial threshold for the CGI allowing the occurrence of a constituted post-traumatic stress disorder to be predicted, defined by a score greater than or equal to 33 on the PCL5. The objective is to set up a systematic recall protocol for subjects presenting with a state of acute stress for which an initial CGI score will be higher than the determined threshold, in order to be able, depending on the subsequent symptomatology, to offer early management. and focus of post traumatic stress disorder. This reminder protocol will be integrated into routine practices and deployed on the emergency reception service of Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has experienced a traumatic event in the last 48 hours;
* Patient speaking French;

Exclusion Criteria:

* Patient participating in another clinical trial on the treatment of his psychotraumatic experience.
* Person deprived of liberty (prisoners, defendants);
* Persons under legal protection (protected adults: under guardianship, curatorship, etc.);
* Opposition of the patient to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient who has experienced a traumatic event in the last 48 hours All patients meeting the inclusion criteria will be identified by the staff of the CUMP (medico-psychological emergency unit) either during an intervention (in the emergency department or outside) or during a psychiatric consultation at the emergencies
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Psychometric properties of the CGI as a predictor of occurrence of post-traumatic stress disorder | inclusion
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.)

SECONDARY OUTCOMES:
Correlation between CGI score and Peritraumatic Distress Inventory scale score (PDI) | Inclusion
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of the patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients).
  PDI consists of 13 likert-style items and total score can range from 0 to 52. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Correlation coefficient between CGI score and PCL 5 score at 1 month. | 1 month
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of the patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients).
  The PCL-5 (Post-traumatic stress disorder Checlist version DSM-5) is a self-assessment comprising 20 items that measures the 20 symptoms of a post-traumatic stress disorder from the DSM-5 (MANUAL. DIAGNOSTIC AND STATISTICS. OF DISORDERS MENTALS. 5th edition.).
  The objectives of the PCL-5 are numerous, such as monitoring changes in symptoms during and after treatment, screening individuals with an episode of post-traumatic stress, making a provisional diagnosis.
Correlation coefficient between CGI score and PCL 5 score at 6 months. | 6 months
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of the patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients).
  The PCL-5 (Post-traumatic stress disorder Checlist version DSM-5) is a self-assessment comprising 20 items that measures the 20 symptoms of a post-traumatic stress disorder from the DSM-5 (MANUAL. DIAGNOSTIC AND STATISTICS. OF DISORDERS MENTALS. 5th edition.).
  The objectives of the PCL-5 are numerous, such as monitoring changes in symptoms during and after treatment, screening individuals with an episode of post-traumatic stress, making a provisional diagnosis.
Presence/absence of a major depressive episode at 1 month in connection with traumatic event | 1 month
  Presence/absence of a major depressive episode assessed by the MINI at 1 month. Search for an association between the CGI score and the presence of a major depressive episode.
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.
Presence/absence of a major depressive episode at 6 months in connection with traumatic event | 6 months
  Presence/absence of a major depressive episode assessed by the MINI at 6 month. Search for an association between the CGI score and the presence of a major depressive episode.
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.
Presence/absence of a consumption of alcohol at 1 month in connection with traumatic event | 1 month
  Presence/absence of a consumption of alcohol assessed by the MINI at 1 month. Search for an association between the CGI score and the presence of a consumption of alcohol.
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.
Presence/absence of a consumption of alcohol at 6 months in connection with traumatic event | 6 months
  Presence/absence of a consumption of alcohol assessed by the MINI at 6 month. Search for an association between the CGI score and the presence of a consumption of alcohol.
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.
Presence/absence of a consumption of substances (except alcohol) at 1 month in connection with traumatic event | 1 month
  Presence/absence of a consumption of substances (except alcohol) assessed by the MINI at 1 month. Search for an association between the CGI score and the presence of a consumption of substances (except alcohol).
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.
Presence/absence of a consumption of substances (except alcohol) 6 months in connection with traumatic event | 6 months
  Presence/absence of a consumption of substances (except alcohol) assessed by the MINI at 6 month. Search for an association between the CGI score and the presence of a consumption of substances (except alcohol).
  Mini International Neuropsychiatric Interview (MINI) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Arras General Hospital, Arras
  - Douai General Hospital, Douai
  - Lens General Hospital, Lens
  - Lille University Hospital, Lille

REFERENCES:
- [Background] Vaiva G, Jehel L, Cottencin O, Ducrocq F, Duchet C, Omnes C, Genest P, Rouillon F, Roelandt JL. [Prevalence of trauma-related disorders in the French WHO study: Sante mentale en population generale (SMPG)]. Encephale. 2008 Dec;34(6):577-83. doi: 10.1016/j.encep.2007.11.006. Epub 2008 Apr 2. French. PMID 19081454
- [Background] Kilpatrick DG. The DSM-5 got PTSD right: comment on Friedman (2013). J Trauma Stress. 2013 Oct;26(5):563-6. doi: 10.1002/jts.21844. PMID 24151004
- [Background] Pietrzak RH, Goldstein RB, Southwick SM, Grant BF. Prevalence and Axis I comorbidity of full and partial posttraumatic stress disorder in the United States: results from Wave 2 of the National Epidemiologic Survey on Alcohol and Related Conditions. J Anxiety Disord. 2011 Apr;25(3):456-65. doi: 10.1016/j.janxdis.2010.11.010. Epub 2010 Nov 26. PMID 21168991
- [Background] Vance MC, Kovachy B, Dong M, Bui E. Peritraumatic distress: A review and synthesis of 15 years of research. J Clin Psychol. 2018 Sep;74(9):1457-1484. doi: 10.1002/jclp.22612. Epub 2018 Mar 15. PMID 29543336
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- See also: La CUMP au-delà de l'évènement : rappel téléphonique des rapatriés du Liban, 2006 — https://santepsy.ascodocpsy.org/index.php?lvl=notice_display&id=151378
- See also: Quand traiter le psychotraumatisme ? — https://www.psychiaclic.fr/media/pages/ressources/quand-traiter-le-psychotraumatisme/9fafc8fa72-1633341136/vaiva-quand-traiter-psychotrauma-lpm-2008.pdf